CLINICAL TRIAL: NCT02289729
Title: Study on Patient- and Caregiver-reported Symptoms and Outcomes With Levodopa/Carbidopa Intestinal Gel for the Treatment of Advanced Parkinson's Disease
Brief Title: Patient- and Caregiver-reported Symptoms and Outcomes With Levodopa/Carbidopa Intestinal Gel for the Treatment of Advanced Parkinson's Disease
Acronym: ADEQUA
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P14-335
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2017-11

CONDITIONS: Parkinson's Disease
Keywords: Duodopa; Advanced Parkinson's Disease; Levodopa/Carbidopa intestinal gel
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Levodopa/carbidopa intestinal gel (LCIG) prescribed in the usual manner, in accordance with the terms of the local marketing authorization, for participants with advanced Parkinson's disease with motor fluctuation not well responding to conventional therapies.

SUMMARY:
Patient reported outcomes (PRO) have become an important endpoint assessed in clinical trials. It is important to understand the relationship between medication and patients' symptomatology, quality of life and well-being. We predict levodopa/carbidopa intestinal gel (LCIG; Duodopa) will significantly improve quality of life and emotional well-being compared to baseline in patients with advance Parkinson disease (APD) not well controlled with conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced levodopa-responsive Parkinson's disease, with at least, 2 hours "off" time or 2 hours of dyskinesia based on clinician's/investigator's medical judgment
* Patients with advanced Parkinson's disease with severe motor fluctuations and dyskinesia when combination of conventional PD treatments was unable to satisfactory control symptoms.
* Patients with advanced Parkinson's disease who meet the criteria for use of Levodopa/Carbidopa Intestinal Gel (LCIG) established in the summary of product characteristics, Spanish Neurology Society (SEN) guidelines, local/regional directories (CCAA) or site's protocols for use of LCIG in common clinical practice.
* The decision to treat with LCIG is made by the physician prior to any decision to approach the patient to participate in this study.
* Patients with a cognitive level enough to complete the questionnaires, confirmed by a Mini-mental state examination (MMSE) score of at least 26 points, according to the recommendation of the Movement Disorder Society (MDS) task force on dementia in Parkinson's Disease (PD)

Exclusion Criteria:

* LCIG's contraindications included in the Summary of Product Characteristics (product label)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced Parkinson's Disease patients
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2014-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesc Valldeoriola, MD, Principal Investigator — Hospital Clinic of Barcelona

REFERENCES:
- [Derived] Wetmore JB, Arbelo JM, Catalan MJ, Valldeoriola F, Rodriguez-Blazquez C, Martinez-Martin P. Psychometric Properties of the Apathy Scale in Advanced Parkinson's Disease. Parkinsons Dis. 2019 Mar 28;2019:1965394. doi: 10.1155/2019/1965394. eCollection 2019. PMID 31031906

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 62 participants were enrolled; 59 were evaluable and 3 were non-evaluable because they did not participate in the nasoduodenal test phase and they did not receive any dose of levodopa/carbidopa intestinal infusion gel (LCIG).
Groups:
- All Participants: LCIG prescribed in the usual manner, in accordance with the terms of the local marketing authorization, for participants with advanced Parkinson's disease with motor fluctuation not well responding to conventional therapies.
Period: Overall Study
Arm/Group | All Participants
Started | 59
Completed | 53
Not Completed | 6
Not completed — Lack of Efficacy | 3
Not completed — Very Narrow Therapeutic Margin | 1
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: participants who received at least 1 dose of LCIG
Arm/Group | All Participants
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.93 (7.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Parkinson's Disease Questionnaire-39 Item (PDQ-39) Global Score at Month 6
Description: The PDQ-39 contains 39 items: mobility (items 1-10), activities of daily living (items 11-16), emotional well-being (items 17-22), stigma (items 23-26), social support (items 27-29), cognitions (items 30-33), communication (items 34-36), and bodily discomfort (items 37-39). Participants are asked to indicate the frequency of each event by selecting one of 5 options (score 0 to 4 on a Likert scale). The global score was calculated by expressing summed item scores as a percentage score ranging between 0 and 100. The lower scores indicate a better perceived health status and higher scores are associated with more health problems.
Time Frame: Baseline, Month 6 (±15 days)
Population: Intent-to-Treat population: participants who received at least one dose of the study medication (LCIG) and completed baseline and end-of-treatment assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | -12.81 (14.65)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 0.0001, t-test

2. Primary Outcome: Change From Baseline in PDQ-39 Mobility Domain Score at Month 6
Description: The PDQ-39 contains 39 items grouped in 8 domains: mobility (items 1-10), activities of daily living (items 11-16), emotional well-being (items 17-22), stigma (items 23-26), social support (items 27-29), cognitions (items 30-33), communication (items 34-36), and bodily discomfort (items 37-39). Participants are asked to indicate the frequency of each event by selecting one of 5 options (Likert scale): never, occasionally, sometimes, often, always or cannot do at all, scoring 0, 1, 2, 3 or 4, respectively. The mobility domain score was calculated by expressing summed item scores as a percentage score ranging between 0 and 100. The lower scores indicate a better perceived health status and higher scores are associated with more health problems.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | -16.92 (24.90)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 0.0001, t-test

3. Primary Outcome: Change From Baseline in PDQ-39 Activities of Daily Living Domain Score at Month 6
Description: The PDQ-39 contains 39 items grouped in 8 domains: mobility (items 1-10), activities of daily living (items 11-16), emotional well-being (items 17-22), stigma (items 23-26), social support (items 27-29), cognitions (items 30-33), communication (items 34-36), and bodily discomfort (items 37-39). Participants are asked to indicate the frequency of each event by selecting one of 5 options (Likert scale): never, occasionally, sometimes, often, always or cannot do at all, scoring 0, 1, 2, 3 or 4, respectively. The activities of daily living domain score was calculated by expressing summed item scores as a percentage score ranging between 0 and 100. The lower scores indicate a better perceived health status and higher scores are associated with more health problems.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | -18.43 (23.52)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 0.0001, t-test

4. Primary Outcome: Change From Baseline in PDQ-39 Emotional Well-Being Domain Score at Month 6
Description: The PDQ-39 contains 39 items grouped in 8 domains: mobility (items 1-10), activities of daily living (items 11-16), emotional well-being (items 17-22), stigma (items 23-26), social support (items 27-29), cognitions (items 30-33), communication (items 34-36), and bodily discomfort (items 37-39). Participants are asked to indicate the frequency of each event by selecting one of 5 options (Likert scale): never, occasionally, sometimes, often, always or cannot do at all, scoring 0, 1, 2, 3 or 4, respectively. The emotional well-being domain score was calculated by expressing summed item scores as a percentage score ranging between 0 and 100. The lower scores indicate a better perceived health status and higher scores are associated with more health problems.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | -13.06 (19.56)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 0.0001, t-test

5. Primary Outcome: Change From Baseline in PDQ-39 Stigma Domain Score at Month 6
Description: The PDQ-39 contains 39 items grouped in 8 domains: mobility (items 1-10), activities of daily living (items 11-16), emotional well-being (items 17-22), stigma (items 23-26), social support (items 27-29), cognitions (items 30-33), communication (items 34-36), and bodily discomfort (items 37-39). Participants are asked to indicate the frequency of each event by selecting one of 5 options (Likert scale): never, occasionally, sometimes, often, always or cannot do at all, scoring 0, 1, 2, 3 or 4, respectively. The stigma domain score was calculated by expressing summed item scores as a percentage score ranging between 0 and 100. The lower scores indicate a better perceived health status and higher scores are associated with more health problems.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | -6.85 (20.53)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.0328, t-test

6. Primary Outcome: Change From Baseline in PDQ-39 Social Support Domain Score at Month 6
Description: The PDQ-39 contains 39 items grouped in 8 domains: mobility (items 1-10), activities of daily living (items 11-16), emotional well-being (items 17-22), stigma (items 23-26), social support (items 27-29), cognitions (items 30-33), communication (items 34-36), and bodily discomfort (items 37-39). Participants are asked to indicate the frequency of each event by selecting one of 5 options (Likert scale): never, occasionally, sometimes, often, always or cannot do at all, scoring 0, 1, 2, 3 or 4, respectively. The social support domain score was calculated by expressing summed item scores as a percentage score ranging between 0 and 100. The lower scores indicate a better perceived health status and higher scores are associated with more health problems.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | -2.08 (15.56)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.4183, t-test

7. Primary Outcome: Change From Baseline in PDQ-39 Cognition Domain Score at Month 6
Description: The PDQ-39 contains 39 items grouped in 8 domains: mobility (items 1-10), activities of daily living (items 11-16), emotional well-being (items 17-22), stigma (items 23-26), social support (items 27-29), cognitions (items 30-33), communication (items 34-36), and bodily discomfort (items 37-39). Participants are asked to indicate the frequency of each event by selecting one of 5 options (Likert scale): never, occasionally, sometimes, often, always or cannot do at all, scoring 0, 1, 2, 3 or 4, respectively. The cognition domain score was calculated by expressing summed item scores as a percentage score ranging between 0 and 100. The lower scores indicate a better perceived health status and higher scores are associated with more health problems.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | -13.22 (19.94)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 0.0001, t-test

8. Primary Outcome: Change From Baseline in PDQ-39 Communication Domain Score at Month 6
Description: The PDQ-39 contains 39 items grouped in 8 domains: mobility (items 1-10), activities of daily living (items 11-16), emotional well-being (items 17-22), stigma (items 23-26), social support (items 27-29), cognitions (items 30-33), communication (items 34-36), and bodily discomfort (items 37-39). Participants are asked to indicate the frequency of each event by selecting one of 5 options (Likert scale): never, occasionally, sometimes, often, always or cannot do at all, scoring 0, 1, 2, 3 or 4, respectively. The communication domain score was calculated by expressing summed item scores as a percentage score ranging between 0 and 100. The lower scores indicate a better perceived health status and higher scores are associated with more health problems.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | -9.13 (17.17)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.0003, t-test

9. Primary Outcome: Change From Baseline in PDQ-39 Bodily Discomfort Domain Score at Month 6
Description: The PDQ-39 contains 39 items grouped in 8 domains: mobility (items 1-10), activities of daily living (items 11-16), emotional well-being (items 17-22), stigma (items 23-26), social support (items 27-29), cognitions (items 30-33), communication (items 34-36), and bodily discomfort (items 37-39). Participants are asked to indicate the frequency of each event by selecting one of 5 options (Likert scale): never, occasionally, sometimes, often, always or cannot do at all, scoring 0, 1, 2, 3 or 4, respectively. The bodily discomfort domain score was calculated by expressing summed item scores as a percentage score ranging between 0 and 100. The lower scores indicate a better perceived health status and higher scores are associated with more health problems.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | -9.13 (24.93)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.0109, t-test

10. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale Part III (UPDRS-III): Motor Examination at Month 6
Description: The UPDRS is an investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The UPDRS-III was used in ON state. The motor examination contains 27 items. Each item is scored in a Likert scale from 0 to 4. The UPDRS-III score was calculated summing the score of each item, ranging from 0 to 108, with higher score indicating more impairment.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 53
units on a scale | -6.51 (11.83)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.0002, t-test

11. Secondary Outcome: Change From Baseline in the Non-Motor Symptom Scale (NMSS) Global Score at Month 6
Description: The NMSS measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular including falls (items 1-2), sleep/fatigue (items 3-6), mood/cognition (items 7-12), perceptual problems/hallucinations (items 13-15), attention/memory (items 16-18), gastrointestinal tract (items 19-21), urinary (items 22-24), sexual function (items 25-26), and miscellaneous (pain, taste/smell, weight change, excessive sweating; items 27-30). Severity is rated on a scale from 0 (none) to 3 (severe) and frequency is rated on a scale from 1 (rarely) to 4 (very frequent). The global score was calculated summing the score of each item (severity x frequency), ranging from 0 to 360, with a lower score indicating fewer symptoms. A negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | -35.75 (31.12)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 0.0001, t-test

12. Secondary Outcome: Change From Baseline in NMSS Cardiovascular Domain Score at Month 6
Description: The NMSS measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular including falls (items 1-2), sleep/fatigue (items 3-6), mood/cognition (items 7-12), perceptual problems/hallucinations (items 13-15), attention/memory (items 16-18), gastrointestinal tract (items 19-21), urinary (items 22-24), sexual function (items 25-26), and miscellaneous (pain, taste/smell, weight change, excessive sweating; items 27-30). Severity is rated on a scale from 0 (none) to 3 (severe) and frequency is rated on a scale from 1 (rarely) to 4 (very frequent). The cardiovascular domain score ranges from 0 to 24 with a lower score indicating fewer symptoms. A negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | -1.81 (3.51)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.0002, signed-rank test

13. Secondary Outcome: Change From Baseline in NMSS Sleep/Fatigue Domain Score at Month 6
Description: The NMSS measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular including falls (items 1-2), sleep/fatigue (items 3-6), mood/cognition (items 7-12), perceptual problems/hallucinations (items 13-15), attention/memory (items 16-18), gastrointestinal tract (items 19-21), urinary (items 22-24), sexual function (items 25-26), and miscellaneous (pain, taste/smell, weight change, excessive sweating; items 27-30). Severity is rated on a scale from 0 (none) to 3 (severe) and frequency is rated on a scale from 1 (rarely) to 4 (very frequent). The sleep/fatigue domain score ranges from 0 to 48 with a lower score indicating fewer symptoms. A negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | -8.73 (7.77)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 0.0001, t-test

14. Secondary Outcome: Change From Baseline in NMSS Mood/Cognition Domain Score at Month 6
Description: The NMSS measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular including falls (items 1-2), sleep/fatigue (items 3-6), mood/cognition (items 7-12), perceptual problems/hallucinations (items 13-15), attention/memory (items 16-18), gastrointestinal tract (items 19-21), urinary (items 22-24), sexual function (items 25-26), and miscellaneous (pain, taste/smell, weight change, excessive sweating; items 27-30). Severity is rated on a scale from 0 (none) to 3 (severe) and frequency is rated on a scale from 1 (rarely) to 4 (very frequent). The mood/cognition domain score ranges from 0 to 72 with a lower score indicating fewer symptoms. A negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | -5.83 (13.84)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.0038, t-test

15. Secondary Outcome: Change From Baseline in NMSS Perceptual Problems/Hallucinations Domain Score at Month 6
Description: The NMSS measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular including falls (items 1-2), sleep/fatigue (items 3-6), mood/cognition (items 7-12), perceptual problems/hallucinations (items 13-15), attention/memory (items 16-18), gastrointestinal tract (items 19-21), urinary (items 22-24), sexual function (items 25-26), and miscellaneous (pain, taste/smell, weight change, excessive sweating; items 27-30). Severity is rated on a scale from 0 (none) to 3 (severe) and frequency is rated on a scale from 1 (rarely) to 4 (very frequent). The perceptual problems/hallucinations domain score ranges from 0 to 36 with a lower score indicating fewer symptoms. A negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | 2.12 (5.03)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 0.0001, signed-rank test

16. Secondary Outcome: Change From Baseline in NMSS Attention/Memory Domain Score at Month 6
Description: The NMSS measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular including falls (items 1-2), sleep/fatigue (items 3-6), mood/cognition (items 7-12), perceptual problems/hallucinations (items 13-15), attention/memory (items 16-18), gastrointestinal tract (items 19-21), urinary (items 22-24), sexual function (items 25-26), and miscellaneous (pain, taste/smell, weight change, excessive sweating; items 27-30). Severity is rated on a scale from 0 (none) to 3 (severe) and frequency is rated on a scale from 1 (rarely) to 4 (very frequent). The attention/memory domain score ranges from 0 to 36 with a lower score indicating fewer symptoms. A negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | -1.12 (6.21)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.0274, signed-rank test

17. Secondary Outcome: Change From Baseline in NMSS Gastrointestinal Tract Domain Score at Month 6
Description: The NMSS measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular including falls (items 1-2), sleep/fatigue (items 3-6), mood/cognition (items 7-12), perceptual problems/hallucinations (items 13-15), attention/memory (items 16-18), gastrointestinal tract (items 19-21), urinary (items 22-24), sexual function (items 25-26), and miscellaneous (pain, taste/smell, weight change, excessive sweating; items 27-30). Severity is rated on a scale from 0 (none) to 3 (severe) and frequency is rated on a scale from 1 (rarely) to 4 (very frequent). The gastrointestinal tract domain score ranges from 0 to 36 with a lower score indicating fewer symptoms; a negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | -3.58 (5.08)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 0.0001, signed-rank test

18. Secondary Outcome: Change From Baseline in NMSS Urinary Domain Score at Month 6
Description: The NMSS measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular including falls (items 1-2), sleep/fatigue (items 3-6), mood/cognition (items 7-12), perceptual problems/hallucinations (items 13-15), attention/memory (items 16-18), gastrointestinal tract (items 19-21), urinary (items 22-24), sexual function (items 25-26), and miscellaneous (pain, taste/smell, weight change, excessive sweating; items 27-30). Severity is rated on a scale from 0 (none) to 3 (severe) and frequency is rated on a scale from 1 (rarely) to 4 (very frequent). The urinary domain score ranges from 0 to 36 with a lower score indicating fewer symptoms.A negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | -5.19 (10.24)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.0006, t-test

19. Secondary Outcome: Change From Baseline in NMSS Sexual Function Domain Score at Month 6
Description: The NMSS measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular including falls (items 1-2), sleep/fatigue (items 3-6), mood/cognition (items 7-12), perceptual problems/hallucinations (items 13-15), attention/memory (items 16-18), gastrointestinal tract (items 19-21), urinary (items 22-24), sexual function (items 25-26), and miscellaneous (pain, taste/smell, weight change, excessive sweating; items 27-30). Severity is rated on a scale from 0 (none) to 3 (severe) and frequency is rated on a scale from 1 (rarely) to 4 (very frequent). The sexual function domain score ranges from 0 to 24 with a lower score indicating fewer symptoms. A negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | -2.94 (6.80)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.0010, signed-rank test

20. Secondary Outcome: Change From Baseline in NMSS Miscellaneous Domain Score at Month 6
Description: The NMSS measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular including falls (items 1-2), sleep/fatigue (items 3-6), mood/cognition (items 7-12), perceptual problems/hallucinations (items 13-15), attention/memory (items 16-18), gastrointestinal tract (items 19-21), urinary (items 22-24), sexual function (items 25-26), and miscellaneous (pain, taste/smell, weight change, excessive sweating; items 27-30). Severity is rated on a scale from 0 (none) to 3 (severe) and frequency is rated on a scale from 1 (rarely) to 4 (very frequent). The miscellaneous domain score ranges from 0 to 48 with a lower score indicating fewer symptoms. A negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 51
units on a scale | -4.47 (8.00)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.0002, t-test

21. Secondary Outcome: Change From Baseline in the Norris/Bond-Lader Visual Analogue Scale (VAS) Mean Global Score at Month 6
Description: The Norris/Bond-Lader VAS measures emotional well-being status with a 16-item visual analogue mood rating scale. The VAS consisted of 16 visual analogue items each representing opposite extremes of mood, with the following labels at each end: alert/drowsy, calm/excited, strong/weak, muzzy/clear-headed, well-coordinated/clumsy, lethargic/energetic, contented/dreamy, incompetent/proficient, happy/sad, antagonistic/amicable, interested/bored, withdrawn/gregarious. These scales loaded on 3 domains (alert, strong, clear-headed, well-coordinated, energetic, quick-witted, attentive, proficient, interested); (contented, tranquil, happy, amicable, gregarious); (calm, relaxed). For each individual scale, a line was drawn between each mood state and its opposite and participants rated their current mood by placing a vertical mark on the line. Scores (global, and for each domain) ranged from 0 to 100, with lower scores indicating more positive mood.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 51
units on a scale | -6.63 (21.15)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.0297, t-test

22. Secondary Outcome: Change From Baseline in the Norris/Bond-Lader Visual Analogue Scale (VAS) Alertness/Sedation Sub-Scale Score at Month 6
Description: as for outcome 21
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 51
units on a scale | -7.38 (23.27)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.0279, t-test

23. Secondary Outcome: Change From Baseline in the Norris/Bond-Lader Visual Analogue Scale (VAS) Contented/Discontented Sub-Scale Score at Month 6
Description: as for outcome 21
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 51
units on a scale | -3.37 (21.92)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.2777, t-test

24. Secondary Outcome: Change From Baseline in the Norris/Bond-Lader Visual Analogue Scale (VAS) Calmness/Relaxation Sub-Scale Score at Month 6
Description: as for outcome 21
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 51
units on a scale | -11.58 (27.94)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.0047, t-test

25. Secondary Outcome: Change From Baseline in Parkinson Fatigue Scale (PFS-16) at Month 6
Description: The PFS-16 comprises 16 items with five polytomous response categories (strongly disagree, disagree, do not agree or disagree, agree, and strongly agree). Responses were scored from 0 (strongly disagree) to 4 (strongly agree), yielding a summed total score ranging from 0 (no fatigue) to 64 (most severe fatigue). The cut-point of ≥ 3.30 was used to identified those perceiving fatigue to be a problem.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 51
units on a scale | -0.56 (1.01)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.0003, t-test

26. Secondary Outcome: Change From Baseline in the Score of the Apathy Scale (AS) to Month 6
Description: The AS is an inventory of 14 questions that assess cognitive and behavioral symptoms of emotional apathy. Each is rated from 0 to 3 on a Likert scale. The total scores for AS ranges from 0 (no apathy) to 42 (most apathetic). AS scores ≥ 14 were considered apathetic.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | -0.52 (6.86)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 0.5877, t-test

27. Secondary Outcome: Change From Baseline in Beck Depression Inventory, Second Edition (BDI-II) at Month 6
Description: The BDI-II is a 21-item self-report multiple-choice inventory. Items are rated on a 4-point scale ranging from 0 to 3 based on severity of each item. The maximum total score is 63. Raw scores from 0-13 indicates minimal depression, 14-19 indicates mild depression, 20-28 indicates moderate depression, and 29-63 indicates severe depression.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | -5.15 (9.39)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.0002, t-test

28. Secondary Outcome: Change From Baseline in Beck Anxiety Inventory (BAI) at Month 6
Description: The BAI is a 21-item self-report multiple-choice inventory. Items are rated on a 4-point scale ranging from 0 to 3 based on severity of each item. The maximum total score is 63. Raw scores from 0-7 indicates minimal anxiety, 8-15 indicates mild anxiety, 16-25 indicates moderate anxiety, and 25-63 indicates severe anxiety.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | -6.21 (9.57)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 0.0001, t-test

29. Secondary Outcome: Change From Baseline in the Treatment Satisfaction With Medicines Questionnaire (SATMED-Q) Composite Score at Month 6
Description: The SATMED-Q is a 17-item questionnaire. Items are grouped in 6 domains: undesirable side effects (items 1-3), treatment effectiveness (items 4-6), convenience of use (items 7-9), impact on daily living activities (items 10-12), medical care (items 13-14), and global satisfaction (items 15-17). Items are rated on a 5-point scale ranging from 0 to 4. Summing up the direct scores of the items yields a total composite score ranging between 0 and 68, which was transformed to a minimum of 0 (most satisfied) and a maximum of 100 (least satisfied).
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | 16.15 (16.80)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 0.0001, t-test

30. Secondary Outcome: Change From Baseline in the Treatment Satisfaction With Medicines Questionnaire (SATMED-Q) Undesirable Side Effects at Month 6
Description: The SATMED-Q is a 17-item questionnaire. Items are grouped in 6 domains: undesirable side effects (items 1-3), treatment effectiveness (items 4-6), convenience of use (items 7-9), impact on daily living activities (items 10-12), medical care (items 13-14), and global satisfaction (items 15-17). Items are rated on a 4-point scale ranging from 0 to 4. Summing up the direct scores of the items yields a total undesirable side effects score ranging between 0 and 12, which was transformed to a minimum of 0 (most satisfied) and a maximum of 100 (least satisfied).
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 46
units on a scale | -25.00 (39.05)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 0.0001, signed-rank test

31. Secondary Outcome: Change From Baseline in the Treatment Satisfaction With Medicines Questionnaire (SATMED-Q) Treatment Effectiveness at Month 6
Description: The SATMED-Q is a 17-item questionnaire. Items are grouped in 6 domains: undesirable side effects (items 1-3), treatment effectiveness (items 4-6), convenience of use (items 7-9), impact on daily living activities (items 10-12), medical care (items 13-14), and global satisfaction (items 15-17). Items are rated on a 4-point scale ranging from 0 to 4. Summing up the direct scores of the items yields a total treatment effectiveness score ranging between 0 and 12, which was transformed to a minimum of 0 (most satisfied) and a maximum of 100 (least satisfied).
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 51
units on a scale | 30.39 (31.57)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 0.0001, t-test

32. Secondary Outcome: Change From Baseline in the Treatment Satisfaction With Medicines Questionnaire (SATMED-Q) Convenience of Use at Month 6
Description: The SATMED-Q is a 17-item questionnaire. Items are grouped in 6 domains: undesirable side effects (items 1-3), treatment effectiveness (items 4-6), convenience of use (items 7-9), impact on daily living activities (items 10-12), medical care (items 13-14), and global satisfaction (items 15-17). Items are rated on a 4-point scale ranging from 0 to 4. Summing up the direct scores of the items yields a total convenience of use score ranging between 0 and 12, which was transformed to a minimum of 0 (most satisfied) and a maximum of 100 (least satisfied).
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 51
units on a scale | 19.77 (33.83)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.0001, t-test

33. Secondary Outcome: Change From Baseline in the Treatment Satisfaction With Medicines Questionnaire (SATMED-Q) Impact on Daily Living Activities at Month 6
Description: The SATMED-Q is a 17-item questionnaire. Items are grouped in 6 domains: undesirable side effects (items 1-3), treatment effectiveness (items 4-6), convenience of use (items 7-9), impact on daily living activities (items 10-12), medical care (items 13-14), and global satisfaction (items 15-17). Items are rated on a 4-point scale ranging from 0 to 4. Summing up the direct scores of the items yields a total impact on daily living activities score ranging between 0 and 12, which was transformed to a minimum of 0 (most satisfied) and a maximum of 100 (least satisfied).
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | 18.75 (30.78)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 0.0001, signed-rank test

34. Secondary Outcome: Change From Baseline in the Treatment Satisfaction With Medicines Questionnaire (SATMED-Q) Medical Care at Month 6
Description: The SATMED-Q is a 17-item questionnaire. Items are grouped in 6 domains: undesirable side effects (items 1-3), treatment effectiveness (items 4-6), convenience of use (items 7-9), impact on daily living activities (items 10-12), medical care (items 13-14), and global satisfaction (items 15-17). Items are rated on a 4-point scale ranging from 0 to 4. Summing up the direct scores of the items yields a total medical care score ranging between 0 and 8, which was transformed to a minimum of 0 (most satisfied) and a maximum of 100 (least satisfied).
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 52
units on a scale | 4.09 (22.51)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.2428, signed-rank test

35. Secondary Outcome: Change From Baseline in the Treatment Satisfaction With Medicines Questionnaire (SATMED-Q) Global Satisfaction at Month 6
Description: The SATMED-Q is a 17-item questionnaire. Items are grouped in 6 domains: undesirable side effects (items 1-3), treatment effectiveness (items 4-6), convenience of use (items 7-9), impact on daily living activities (items 10-12), medical care (items 13-14), and global satisfaction (items 15-17). Items are rated on a 4-point scale ranging from 0 to 4. Summing up the direct scores of the items yields a total global satisfaction score ranging between 0 and 12, which was transformed to a minimum of 0 (most satisfied) and a maximum of 100 (least satisfied).
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 51
units on a scale | 44.44 (32.00)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.0687, t-test

36. Secondary Outcome: Change From Baseline in the Scale of Quality of Life of Caregivers (SQLC) Composite Score at Month 6
Description: The SQLC is designed to both qualitatively and quantitatively evaluate the impact of a patient's disease on the caregiver's quality of life. The SQLC questionnaire consists of 16 questions that evaluate 3 domains: professional activities (questions 1-4), social and leisure activities (questions 5-9), and caregiving responsibilities (questions 10-16). Composite scores range from 0 to 149, with higher scores indicating higher quality of life.
Time Frame: Baseline, Month 6 (±15 days)
Population: Intent-to-Treat population: participants (and caregivers) who received at least one dose of the study medication (LCIG) and completed baseline and end-of-treatment assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 47
units on a scale | 3.21 (21.57)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.3126, t-test

37. Secondary Outcome: Change From Baseline in the Scale of Quality of Life of Caregivers (SQLC) Professional Activities at Month 6
Description: The SQLC is designed to both qualitatively and quantitatively evaluate the impact of a patient's disease on the caregiver's quality of life. The SQLC questionnaire consists of 16 questions that evaluate 3 domains: professional activities (questions 1-4), social and leisure activities (questions 5-9), and caregiving responsibilities (questions 10-16). Professional activities scores range from 0 to 38, with higher scores indicating higher quality of life.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 47
units on a scale | 2.55 (12.06)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.1533, t-test

38. Secondary Outcome: Change From Baseline in the Scale of Quality of Life of Caregivers (SQLC) Social and Leisure Activities at Month 6
Description: The SQLC is designed to both qualitatively and quantitatively evaluate the impact of a patient's disease on the caregiver's quality of life. The SQLC questionnaire consists of 16 questions that evaluate 3 domains: professional activities (questions 1-4), social and leisure activities (questions 5-9), and caregiving responsibilities (questions 10-16). Social and leisure activities scores range from 0 to 58, with higher scores indicating higher quality of life.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 47
units on a scale | -0.21 (6.18)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.8145, t-test

39. Secondary Outcome: Change From Baseline in the Scale of Quality of Life of Caregivers (SQLC) Caregiving Responsibilities at Month 6
Description: The SQLC is designed to both qualitatively and quantitatively evaluate the impact of a patient's disease on the caregiver's quality of life. The SQLC questionnaire consists of 16 questions that evaluate 3 domains: professional activities (questions 1-4), social and leisure activities (questions 5-9), and caregiving responsibilities (questions 10-16). Caregiving responsibilities scores range from 0 to 53, with higher scores indicating higher quality of life.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 47
units on a scale | 0.87 (7.11)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.4048, t-test

40. Secondary Outcome: Change From Baseline in Zarit Burden Interview (ZBI) at Month 6
Description: The ZBI is a 22-item questionnaire in which caregivers must evaluate the level of agreement on a 5-point Likert scale from 0 to 4. The total score is obtained by the sum of the scores of the items. This total score represents a level of caregiver burden, with a range of 0 indicating no burden to 88 indicating completely overloaded.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 47
units on a scale | -0.32 (10.26)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.8321, t-test

41. Secondary Outcome: Change From Baseline in the Caregiver Stress Index (CSI) at Month 6
Description: The CSI is a 13-item questionnaire based on identified common stressors. Answers are in yes/no format. Scoring is 1 point for each "yes" and 0 for each "no". The total score is obtained by the sum of the scores of the items. Minimum score is 0 (no stress) and maximum score is 13 (most stress). A score ≥ 7 indicates a high level of stress.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 47
units on a scale | -0.55 (2.58)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.1945, signed-rank test

42. Secondary Outcome: Change From Baseline in Goldberg Anxiety and Depression Score (GADS): Depression Sub-Scale for Caregivers at Month 6
Description: The GADS is an 18-item self-report symptom inventory made up of two sub-scales, one for the detection of anxiety and another one for the detection of depression. Both sub-scales are composed of 9 questions. Answers are in yes/no format. Scoring is 1 point for each "yes" and 0 for each "no", with a total sub-scale score of 0 (no anxiety/depression) to 9 (worst anxiety/depression). In the Spanish validation of GADS, the cutoff point to consider probable anxiety disorder is 4 and 2 for probable depression.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 10
units on a scale | 0.20 (2.35)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.7937, t-test

43. Secondary Outcome: Change From Baseline in Goldberg Anxiety and Depression Score (GADS): Anxiety Sub-Scale for Caregivers at Month 6
Description: as for outcome 42
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 10
units on a scale | -1.10 (0.99)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.0234, signed-rank test

44. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI) Questionnaire: Mean Percentage of Work Time Missed (Absenteeism) at Month 6
Description: Absenteeism, presented as the mean percentage of work time missed due to caregiving (as reported on the WPAI), and calculated as: 100*number of hours of work missed due to caregiving / (number of hours of work missed due to caregiving + number of hours worked). WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | All Participants
Number analyzed (Participants) | 9
percentage of work time missed | -7.56 (40.68)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.5922, t-test

45. Secondary Outcome: Change From Baseline in WPAI Questionnaire: Mean Percentage of Impairment While Working Due to Caregiving (Presenteeism)
Description: Presenteeism (the extent to which caregiving decreased productivity) is presented as the mean percentage of impairment while working due to caregiving, and calculated as: 100*scale value of question 5 on the WPAI (between 0 and 10) / 10. WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: percentage of work impairment
Arm/Group | All Participants
Number analyzed (Participants) | 9
percentage of work impairment | 0.00 (18.03)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 1.000, t-test

46. Secondary Outcome: Change From Baseline in WPAI Questionnaire: Mean Percentage of Overall Work Productivity Impairment (OWPI) Due to Caregiving
Description: The mean percentage of OWPI due to caregiving (based on the WPAI questionnaire) is presented, calculated as: Absenteeism (%) + extent to which caregiving decreased productivity (%)* [number of hours worked / (number of hours of work missed due to caregiving + number of hours worked)]. WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: percentage of overall work impairment
Arm/Group | All Participants
Number analyzed (Participants) | 9
percentage of overall work impairment | -6.69 (42.34)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.6481, t-test

47. Secondary Outcome: Change From Baseline in WPAI Questionnaire: Mean Percentage of Activity Impairment Due to Caregiving
Description: Activity impairment due to caregiving (the extent to which caregiving affected the ability to perform usual daily activities) is presented as the mean percentage of activity impairment, calculated as 100*scale value of WPAI question 6 (between 0 and 10) / 10. WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity/activity and 100% representing complete impact on productivity/activity.
Time Frame: Baseline, Month 6 (±15 days)
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: percentage of activity impairment
Arm/Group | All Participants
Number analyzed (Participants) | 9
percentage of activity impairment | -3.33 (22.91)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.6741, t-test

48. Secondary Outcome: Correlation Between Participants' Quality of Life (PDQ-39) and Different Questionnaires at Baseline
Description: Spearman correlation statistics were calculated for the quality of life of the participants (Global PDQ-39, see Outcome Measure 1) and the following scales: UPDRS-III (see Outcome Measure 10), UPDRS-IV (see description below), NMSS (see Outcome Measure 11), BAI (see Outcome Measure 28), BDI-III (see Outcome Measure 27), AS (see Outcome Measure 26), PFS (see Outcome Measure 25), Norris Bond-Lader (NBL) Alertness-Sedation (A-S; see Outcome Measure 22), NBL Contented-Discontented (C-D; see Outcome Measure 23), NBL Calm-Relaxed (C-R; see Outcome Measure 24), ZBI (see Outcome Measure 40), GADS-Anxiety (see Outcome Measure 43), and GADS-Depression (see Outcome Measure 42).
  The UPDRS-IV contains 11 items, each scored in a Likert scale from 0 (normal) to 4 (severe); or a 2-point scale (yes/no format), with 1 point for "yes" and 0 for "no." The global score was calculated summing the score of each item, ranging from 0 to 23, where higher scores are associated with more disability.
Time Frame: Baseline
Population: Intent-to-Treat population: participants (and caregivers) who received at least one dose of the study medication (LCIG) and completed baseline assessments.
Measure: Number; unit: correlation coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 58
correlation coefficient
  PDQ-39 with UPDRS-III | 0.27148
  PDQ-39 with UPDRS-IV | 0.07346
  PDQ-39 with NMSS | 0.20994
  PDQ-39 with BAI | 0.28271
  PDQ-39 with BDI-II | 0.46174
  PDQ-39 with AS: number analyzed (Participants) | 57
  PDQ-39 with AS | 0.08846
  PDQ-39 with PFS: number analyzed (Participants) | 57
  PDQ-39 with PFS | 0.33361
  PDQ-39 with NBL A-S: number analyzed (Participants) | 57
  PDQ-39 with NBL A-S | 0.22085
  PDQ-39 with NBL C-D: number analyzed (Participants) | 57
  PDQ-39 with NBL C-D | 0.35742
  PDQ-39 with NBL C-R: number analyzed (Participants) | 57
  PDQ-39 with NBL C-R | 0.00011
  PDQ-39 with ZBI: number analyzed (Participants) | 54
  PDQ-39 with ZBI | -0.35125
  PDQ-39 with GADS-Anxiety: number analyzed (Participants) | 54
  PDQ-39 with GADS-Anxiety | 0.21311
  PDQ-39 with GADS-Depression: number analyzed (Participants) | 28
  PDQ-39 with GADS-Depression | 0.51846
Statistical Analysis 1: Comparison: All Participants; PDQ-39 with UPDRS-III; Test type: Other; p = 0.0389, Fisher's z Transformation; Fisher's z = 0.27846, 95% CI 2-sided [0.014175 to 0.495059]
Statistical Analysis 2: Comparison: All Participants; PDQ-39 with UPDRS-IV; Test type: Other; p = 0.5852, Fisher's z Transformation; Fisher's z = 0.07359, 95% CI 2-sided [-0.188409 to 0.325580]
Statistical Analysis 3: Comparison: All Participants; PDQ-39 with NMSS; Test type: Other; p = 0.1140, Fisher's z Transformation; Fisher's z = 0.21311, 95% CI 2-sided [-0.051127 to 0.444152]
Statistical Analysis 4: Comparison: All Participants; PDQ-39 with BAI; Test type: Other; p = 0.0311, Fisher's z Transformation; Fisher's z = 0.29062, 95% CI 2-sided [0.026334 to 0.504186]
Statistical Analysis 5: Comparison: All Participants; PDQ-39 with BDI-II; Test type: Other; p = 0.0002, Fisher's z Transformation; Fisher's z = 0.49952, 95% CI 2-sided [0.230995 to 0.643312]
Statistical Analysis 6: Comparison: All Participants; PDQ-39 with AS; Test type: Other; p = 0.5146, Fisher's z Transformation; Fisher's z = 0.08869, 95% CI 2-sided [-0.176169 to 0.341163]
Statistical Analysis 7: Comparison: All Participants; PDQ-39 with PFS; Test type: Other; p = 0.0108, Fisher's z Transformation; Fisher's z = 0.34688, 95% CI 2-sided [0.079996 to 0.546657]
Statistical Analysis 8: Comparison: All Participants; PDQ-39 with NBL A-S; Test type: Other; p = 0.0989, Fisher's z Transformation; Fisher's z = 0.22455, 95% CI 2-sided [-0.042139 to 0.455224]
Statistical Analysis 9: Comparison: All Participants; PDQ-39 with NBL C-D; Test type: Other; p = 0.0060, Fisher's z Transformation; Fisher's z = 0.35742, 95% CI 2-sided [0.106797 to 0.565335]
Statistical Analysis 10: Comparison: All Participants; PDQ-39 with NBL C-R; Test type: Other; p = 0.9993, Fisher's z Transformation; Fisher's z = 0.00011, 95% CI 2-sided [-0.260462 to 0.260673]
Statistical Analysis 11: Comparison: All Participants; PDQ-39 with ZBI; Test type: Other; p = 0.0088, Fisher's z Transformation; Fisher's z = -0.36687, 95% CI 2-sided [-0.565795 to -0.092154]
Statistical Analysis 12: Comparison: All Participants; PDQ-39 with Goldberg-Anxiety; Test type: Other; p = 0.1222, Fisher's z Transformation; Fisher's z = 0.21643, 95% CI 2-sided [-0.057959 to 0.454911]
Statistical Analysis 13: Comparison: All Participants; PDQ-39 with Goldberg-Depression; Test type: Other; p = 0.0041, Fisher's z Transformation; Fisher's z = 0.57423, 95% CI 2-sided [0.180247 to 0.747040]

49. Secondary Outcome: Correlation Between Participants' Quality of Life (PDQ-39) and Different Questionnaires at Month 6
Description: as for outcome 48
Time Frame: Month 6 (±15 days)
Population: Intent-to-Treat population: participants (and caregivers) who received at least one dose of the study medication (LCIG) and completed baseline and Month 6 assessments.
Measure: Number; unit: correlation coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 53
correlation coefficient
  PDQ-39 with UPDRS-III | 0.30902
  PDQ-39 with UPDRS-IV | 0.35220
  PDQ-39 with NMSS: number analyzed (Participants) | 52
  PDQ-39 with NMSS | 0.36814
  PDQ-39 with BAI | 0.60620
  PDQ-39 with BDI-II | 0.56325
  PDQ-39 with AS | 0.23657
  PDQ-39 with PFS | 0.58572
  PDQ-39 with NBL A-S | 0.54139
  PDQ-39 with NBL C-D | 0.54140
  PDQ-39 with NBL C-R | 0.38968
  PDQ-39 with ZBI: number analyzed (Participants) | 48
  PDQ-39 with ZBI | -0.32445
  PDQ-39 with GADS-Anxiety: number analyzed (Participants) | 48
  PDQ-39 with GADS-Anxiety | 0.56873
  PDQ-39 with GADS-Depression: number analyzed (Participants) | 15
  PDQ-39 with GADS-Depression | 0.10855
Statistical Analysis 1: Comparison: All Participants; PDQ-39 with UPDRS-III; Test type: Other; p = 0.0239, Fisher's z Transformation; Fisher's z = 0.31946, 95% CI 2-sided [0.042257 to 0.534657]
Statistical Analysis 2: Comparison: All Participants; PDQ-39 with UPDRS-IV; Test type: Other; p = 0.0093, Fisher's z Transformation; Fisher's z = 0.36796, 95% CI 2-sided [0.090528 to 0.568388]
Statistical Analysis 3: Comparison: All Participants; PDQ-39 with NMSS; Test type: Other; p = 0.0069, Fisher's z Transformation; Fisher's z = 0.38627, 95% CI 2-sided [0.105875 to 0.582517]
Statistical Analysis 4: Comparison: All Participants; PDQ-39 with BAI; Test type: Other; p < 0.0001, Fisher's z Transformation; Fisher's z = 0.70289, 95% CI 2-sided [0.401730 to 0.753097]
Statistical Analysis 5: Comparison: All Participants; PDQ-39 with BDI-II; Test type: Other; p < 0.0001, Fisher's z Transformation; Fisher's z = 0.63758, 95% CI 2-sided [0.345567 to 0.723410]
Statistical Analysis 6: Comparison: All Participants; PDQ-39 with AS; Test type: Other; p = 0.0882, Fisher's z Transformation; Fisher's z = 0.24114, 95% CI 2-sided [-0.036024 to 0.476404]
Statistical Analysis 7: Comparison: All Participants; PDQ-39 with PFS; Test type: Other; p < 0.0001, Fisher's z Transformation; Fisher's z = 0.67113, 95% CI 2-sided [0.374757 to 0.739016]
Statistical Analysis 8: Comparison: All Participants; PDQ-39 with NBL A-S; Test type: Other; p < 0.0001, Fisher's z Transformation; Fisher's z = 0.60612, 95% CI 2-sided [0.317572 to 0.708072]
Statistical Analysis 9: Comparison: All Participants; PDQ-39 with NBL C-D; Test type: Other; p < 0.0001, Fisher's z Transformation; Fisher's z = 0.60613, 95% CI 2-sided [0.317580 to 0.708076]
Statistical Analysis 10: Comparison: All Participants; PDQ-39 with NBL C-R; Test type: Other; p = 0.0036, Fisher's z Transformation; Fisher's z = 0.41143, 95% CI 2-sided [0.133445 to 0.597087]
Statistical Analysis 11: Comparison: All Participants; PDQ-39 with ZBI; Test type: Other; p = 0.0239, Fisher's z Transformation; Fisher's z = -0.33661, 95% CI 2-sided [-0.557217 to -0.044411]
Statistical Analysis 12: Comparison: All Participants; PDQ-39 with Goldberg-Anxiety; Test type: Other; p < 0.0001, Fisher's z Transformation; Fisher's z = 0.64565, 95% CI 2-sided [0.339454 to 0.734221]
Statistical Analysis 13: Comparison: All Participants; PDQ-39 with Goldberg-Depression; Test type: Other; p = 0.7058, Fisher's z Transformation; Fisher's z = 0.10898, 95% CI 2-sided [-0.427482 to 0.588111]

50. Secondary Outcome: Correlation Between Caregivers' Quality of Life (SQLC) and Different Questionnaires at Baseline
Description: Spearman correlation statistics were calculated for the quality of life of the caregivers (Global SQLC, see Outcome Measure ) and the following scales: ZBI (see Outcome Measure 40), GADS-Anxiety (see Outcome Measure 43), and GADS-Depression (see Outcome Measure 42), NBL A-S (see Outcome Measure 22), NBL C-D (see Outcome Measure 23), NBL C-R (see Outcome Measure 24), Global PDQ-39 (see Outcome Measure 1), UPDRS-III (see Outcome Measure 10), UPDRS-IV (see description below), and Global NMSS (see Outcome Measure 11).
  The UPDRS-IV contains 11 items, each scored in a Likert scale from 0 (normal) to 4 (severe); or a 2-point scale (yes/no format), with 1 point for "yes" and 0 for "no." The global score was calculated summing the score of each item, ranging from 0 to 23, where higher scores are associated with more disability.
Time Frame: Baseline
Population: as for outcome 48
Measure: Number; unit: correlation coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 54
correlation coefficient
  SQLC with ZBI | -0.51735
  SQLC with GADS-Anxiety: number analyzed (Participants) | 28
  SQLC with GADS-Anxiety | -0.16188
  SQLC with GADS-Depression: number analyzed (Participants) | 25
  SQLC with GADS-Depression | -0.44739
  SQLC with NBL A-S: number analyzed (Participants) | 53
  SQLC with NBL A-S | 0.06318
  SQLC with NBL C-D: number analyzed (Participants) | 53
  SQLC with NBL C-D | 0.17492
  SQLC with NBL C-R: number analyzed (Participants) | 53
  SQLC with NBL C-R | 0.28618
  SQLC with Global PDQ-39 | -0.35125
  SQLC with UPDRS-III | -0.13353
  SQLC with UPDRS-IV | 0.17659
  SQLC with Global NMSS | 0.01625
Statistical Analysis 1: Comparison: All Participants; SQLC with ZBI; Test type: Other; p < 0.0001, Fisher's z Transformation; Fisher's z = -0.57271, 95% CI 2-sided [-0.689585 to -0.289724]
Statistical Analysis 2: Comparison: All Participants; SQLC with Goldberg Anxiety; Test type: Other; p = 0.4142, Fisher's z Transformation; Fisher's z = -0.16332, 95% CI 2-sided [-0.504489 to 0.224771]
Statistical Analysis 3: Comparison: All Participants; SQLC with Goldberg Depression; Test type: Other; p = 0.0239, Fisher's z Transformation; Fisher's z = -0.48143, 95% CI 2-sided [-0.715956 to -0.063481]
Statistical Analysis 4: Comparison: All Participants; SQLC with NBL A-S; Test type: Other; p = 0.6546, Fisher's z Transformation; Fisher's z = 0.06326, 95% CI 2-sided [-0.210715 to 0.327872]
Statistical Analysis 5: Comparison: All Participants; SQLC with NBL C-D; Test type: Other; p = 0.2114, Fisher's z Transformation; Fisher's z = 0.17674, 95% CI 2-sided [-0.100105 to 0.425116]
Statistical Analysis 6: Comparison: All Participants; SQLC with NBL C-R; Test type: Other; p = 0.0374, Fisher's z Transformation; Fisher's z = 0.29440, 95% CI 2-sided [0.017222 to 0.516523]
Statistical Analysis 7: Comparison: All Participants; SQLC with Global PDQ-39; Test type: Other; p = 0.0088, Fisher's z Transformation; Fisher's z = -0.36687, 95% CI 2-sided [-0.565795 to -0.092154]
Statistical Analysis 8: Comparison: All Participants; SQLC with UPDRS-III; Test type: Other; p = 0.3374, Fisher's z Transformation; Fisher's z = -0.13433, 95% CI 2-sided [-0.387439 to 0.139207]
Statistical Analysis 9: Comparison: All Participants; SQLC with UPDRS-IV; Test type: Other; p = 0.2025, Fisher's z Transformation; Fisher's z = 0.17846, 95% CI 2-sided [-0.095693 to 0.424291]
Statistical Analysis 10: Comparison: All Participants; SQLC with Global NMSS; Test type: Other; p = 0.9076, Fisher's z Transformation; Fisher's z = 0.01625, 95% CI 2-sided [-0.252613 to 0.282777]

51. Secondary Outcome: Correlation Between Caregivers' Quality of Life (SQLC) and Different Questionnaires at Month 6
Description: as for outcome 50
Time Frame: Month 6 (±15 days)
Population: Intent-to-Treat population: participants (and caregivers) who received at least one dose of the study medication (LCIG) and completed Month 6 assessments.
Measure: Number; unit: correlation coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 48
correlation coefficient
  SQLC with ZBI | -0.63324
  SQLC with GADS Anxiety: number analyzed (Participants) | 15
  SQLC with GADS Anxiety | 0.17735
  SQLC with GADS Depression: number analyzed (Participants) | 13
  SQLC with GADS Depression | -0.06976
  SQLC with NBL A-S | -0.11015
  SQLC with NBL C-D | 0.00326
  SQLC with NBL C-R | -0.10256
  SQLC with Global PDQ-39 | -0.32445
  SQLC with UPDRS-III | -0.23226
  SQLC with UPDRS-IV | -0.12942
  SQLC with Global NMSS: number analyzed (Participants) | 47
  SQLC with Global NMSS | 0.11635
Statistical Analysis 1: Comparison: All Participants; SQLC with ZBI; Test type: Other; p < 0.0001, Fisher's z Transformation; Fisher's z = -0.74680, 95% CI 2-sided [-0.777482 to -0.425693]
Statistical Analysis 2: Comparison: All Participants; SQLC with Goldberg Anxiety; Test type: Other; p = 0.5347, Fisher's z Transformation; Fisher's z = 0.17924, 95% CI 2-sided [-0.368382 to 0.632178]
Statistical Analysis 3: Comparison: All Participants; SQLC with Goldberg Depression; Test type: Other; p = 0.8251, Fisher's z Transformation; Fisher's z = -0.06987, 95% CI 2-sided [-0.597767 to 0.500464]
Statistical Analysis 4: Comparison: All Participants; SQLC with NBL A-S; Test type: Other; p = 0.4581, Fisher's z transformation; Fisher's z = -0.11060, 95% CI 2-sided [-0.382323 to 0.179601]
Statistical Analysis 5: Comparison: All Participants; SQLC with NBL C-D; Test type: Other; p = 0.9826, Fisher's z Transformation; Fisher's z = 0.00326, 95% CI 2-sided [-0.281136 to 0.287128]
Statistical Analysis 6: Comparison: All Participants; SQLC with NBL C-R; Test type: Other; p = 0.4899, Fisher's z Transformation; Fisher's z = -0.10293, 95% CI 2-sided [-0.375749 to 0.187021]
Statistical Analysis 7: Comparison: All Participants; SQLC with Global PDQ-39; Test type: Other; p = 0.0239, Fisher's z Transformation; Fisher's z = -0.33661, 95% CI 2-sided [-0.557217 to -0.044411]
Statistical Analysis 8: Comparison: All Participants; SQLC with UPDRS-III; Test type: Other; p = 0.1125, Fisher's z Transformation; Fisher's z = -0.23658, 95% CI 2-sided [-0.484427 to 0.055538]
Statistical Analysis 9: Comparison: All Participants; SQLC with UPDRS-IV; Test type: Other; p = 0.3826, Fisher's z Transformation; Fisher's z = -0.13015, 95% CI 2-sided [-0.398887 to 0.160620]
Statistical Analysis 10: Comparison: All Participants; SQLC with Global NMSS; Test type: Other; p = 0.4382, Fisher's z Transformation; Fisher's z = 0.11688, 95% CI 2-sided [-0.176724 to 0.390468]

ADVERSE EVENTS:
Time Frame: Serious adverse events were reported from the time the physician obtained the participant's informed consent until 30 days or 5 half-lives following the intake of the last dose of physician-prescribed treatment. Mean treatment duration was 6.14 ± 1.10 months (median 6.38 months).
Description: Non-serious adverse events were not collected in this observational study, per protocol.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 18/59
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=59)
Acute myocardial infarction (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Femoral hernia incarcerated (Gastrointestinal disorders) | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Pneumoperitoneum (Gastrointestinal disorders) | 4
Infection (Infections and infestations) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Scapula fracture (Injury, poisoning and procedural complications) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 1
Withdrawal syndrome (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.